CLINICAL TRIAL: NCT01362530
Title: A Phase III, Randomized, Double-Blind, Active Comparator-Controlled Clinical Trial, Conducted Under In-House Blinding Conditions, to Examine the Efficacy and Safety of Aprepitant for the Prevention of Chemotherapy-Induced Nausea and Vomiting (CINV) in Pediatric Patients
Brief Title: A Study of the Safety and Efficacy of Aprepitant for the Prevention of Chemotherapy-Induced Nausea and Vomiting (CINV) in Pediatric Participants (MK-0869-208)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 0869-208
Record Dates: First submitted 2011-05-26; First posted 2011-05-30 (Estimated); Results first posted 2014-04-04 (Estimated); Last update posted 2018-09-25 (Actual); Status verified 2018-08

CONDITIONS: Chemotherapy Induced Nausea and Vomiting
MeSH Terms: conditions — Vomiting | interventions — Aprepitant; Suspensions; Ondansetron

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aprepitant Regimen (Experimental): Cycle 1:
  Participants 12 to 17 years of age, Day 1: aprepitant 125 mg capsule orally (PO) + ondansetron, Days 2 to 3: aprepitant 80 mg capsule PO. Participants 6 months to <12 years of age, Day 1: aprepitant powder for suspension (PFS), 3.0 mg/kg (up to 125 mg) + ondansetron, Days 2 to 3: aprepitant PFS, 2.0 mg/kg (up to 80 mg).
  Optional Cycles 2-6:
  Open-label aprepitant administered in the same manner as in Cycle 1.
  Interventions: Drug: Aprepitant 125 mg; Drug: Aprepitant 80 mg; Drug: Aprepitant powder for suspension (PFS); Drug: Ondansetron; Drug: Emetogenic chemotherapy
- Control Regimen (Placebo Comparator): Cycle 1: Participants 12 to 17 years of age, Day 1: matching placebo for aprepitant 125 mg capsule oral (PO) + ondansetron Days 2 to 3: matching placebo for aprepitant 80 mg capsule PO. Participants 6 months to <12 years of age, Day 1: matching placebo PFS: 3.0 mg/kg (up to 125 mg) + ondansetron, Days 2 to 3: matching placebo PFS: 2.0 mg/kg (up to 80 mg). Optional Cycles 2-6: Open-label aprepitant administered in the same manner as in Cycle 1.
  Interventions: Drug: Ondansetron; Drug: Placebo for Aprepitant 125 mg; Drug: Placebo for Aprepitant 80 mg; Drug: Placebo for Aprepitant PFS; Drug: Emetogenic chemotherapy

INTERVENTIONS:
Drug: Aprepitant 125 mg — On the morning of Day 1: one 125 mg capsule PO 60 minutes prior to chemotherapy for participants 12 to 17 years of age
  Other Names: MK-0869, Emend®
  Arms: Aprepitant Regimen
Drug: Aprepitant 80 mg — On the morning of Days 2 and 3: one 80 mg capsule PO for participants 12 to 17 years of age
  Other Names: MK-0869, Emend®
  Arms: Aprepitant Regimen
Drug: Aprepitant powder for suspension (PFS) — On the morning of Day 1: 3.0 mg/kg (up to 125 mg) PO 60 minutes prior to chemotherapy for participants 6 months to <12 years of age. On the morning of Days 2 and 3: 2.0 mg/kg (up to 80 mg) PO 60 minutes prior to chemotherapy (if applicable) for participants 6 months to <12 years of age
  Other Names: MK-0869, Emend®
  Arms: Aprepitant Regimen
Drug: Ondansetron — Day 1: Administered according to product label for pediatric usage or local standard of care
  Other Names: Zofran™
Drug: Placebo for Aprepitant 125 mg — On the morning of Day 1: one 125 mg capsule PO 60 minutes prior to chemotherapy for participants 12 to 17 years of age
  Arms: Control Regimen
Drug: Placebo for Aprepitant 80 mg — On the morning of Days 2 and 3: one 80 mg capsule PO for participants 12 to 17 years of age
  Arms: Control Regimen
Drug: Placebo for Aprepitant PFS — On the morning of Day 1: 3.0 mg/kg (up to 125 mg) PO 60 minutes prior to chemotherapy for participants 6 months to <12 years of age. On the morning of Days 2 and 3: 2.0 mg/kg (up to 80 mg) PO 60 minutes prior to chemotherapy (if applicable) for participants 6 months to <12 years of age
  Arms: Control Regimen
Drug: Emetogenic chemotherapy — Any moderately or highly emetic chemotherapeutic agent such as cyclophosphamide, doxorubicin, methotrexate, carboplatin, cisplatin, irinotecan, carmustine, ifosfamide, and streptozocin, or chemotherapeutics of a lower emetogenicity that were not previously tolerated. No chemotherapeutic agents were specified by the protocol, and many could potentially have been used."

SUMMARY:
This study will compare the safety and efficacy of a three-day oral aprepitant regimen (aprepitant plus ondansetron) to ondansetron alone in the prevention of chemotherapy-induced nausea and vomiting (CINV) in the 120 hours following the initiation of chemotherapy in pediatric participants. Those who complete this first cycle of treatment and meet certain eligibility criteria will have the option of continuing for 5 additional cycles of open-label aprepitant.

ELIGIBILITY:
Inclusion Criteria:

Cycle 1:

* Is 6 months to 17 years of age at time of study entry
* Is scheduled to receive chemotherapeutic agent(s) associated with moderate, high risk or very high risk of vomiting for a documented malignancy, or a chemotherapy regimen not previously tolerated due to vomiting
* Is expected to receive ondansetron as part of their antiemetic regimen
* If female and has begun menses, must has a negative urine pregnancy test prior to

randomization. A female who is of reproductive potential agrees to remain abstinent or use a barrier form of contraception for at least 14 days prior to, throughout, and for at least one month following the last dose of study medication

* If >10 years old, have a Karnofsky score ≥ 60; if ≤ 10 years have a Lansky Play Performance score ≥ 60
* Have a predicted life expectancy of ≥ 3 months

Optional Cycles 2-6:

* Participant has, in the opinion of the investigator, completed the preceding cycle of chemotherapy and related study procedures satisfactorily

Exclusion Criteria:

Cycle 1:

* Has vomited in the 24 hours prior to Treatment Day 1
* Is scheduled to receive stem cell rescue therapy in conjunction with study related course(s) of emetogenic chemotherapy
* Has received or will receive radiation therapy to the abdomen or pelvis within a week prior to Treatment Day 1 or during the course of the study
* Is pregnant or breast feeding
* Is allergic to aprepitant, ondansetron, or any other 5-hydroxytryptamine type-3 receptor (5-HT3) antagonist
* Has a symptomatic primary or metastatic CNS malignancy causing nausea and/or vomiting
* History of QT prolongation or taking other medicinal products that lead to QT prolongation
* Has an active infection (e.g., pneumonia), congestive heart failure, bradyarrhythmia, or any uncontrolled disease (e.g., diabetic ketoacidosis, gastrointestinal obstruction) except for malignancy, which in the opinion of the investigator, might confound the results of the study or pose unwarranted risk in administering study drug to the participant
* Has had benzodiazepine or opioid therapy initiated within 48 hours of study drug administration, except for single daily doses of triazolam, temazepam, or midazolam
* Has been started on systemic corticosteroid therapy within 72 hours prior to study drug administration or is planned to receive a corticosteroid as part of the chemotherapy regimen
* Is currently taking warfarin

Optional Cycles 2-6:

* All exclusion criteria from Cycle 1 apply except for vomiting in the 24 hours prior to Treatment Day 1

Ages: 6 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 307 (Actual)
Dates: Start 2011-09-13 (Actual); Primary Completion 2013-03-14 (Actual); Study Completion 2013-08-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Kang HJ, Loftus S, Taylor A, DiCristina C, Green S, Zwaan CM. Aprepitant for the prevention of chemotherapy-induced nausea and vomiting in children: a randomised, double-blind, phase 3 trial. Lancet Oncol. 2015 Apr;16(4):385-94. doi: 10.1016/S1470-2045(15)70061-6. Epub 2015 Mar 12. PMID 25770814
- [Derived] Kang HJ, Loftus S, DiCristina C, Green S, Pong A, Zwaan CM. Aprepitant for the prevention of chemotherapy-induced nausea and vomiting in paediatric subjects: An analysis by age group. Pediatr Blood Cancer. 2018 Oct;65(10):e27273. doi: 10.1002/pbc.27273. Epub 2018 Jun 12. PMID 29893452
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/study.html?id=0869-208&kw=0869-208&tab=access

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The base study consisted of once cycle of treatment (Cycle 1). Participants in either treatment group who met the eligibility criteria were eligible to participate in optional open-label aprepitant treatment for an additional 5 cycles (Cycles 2-6).
Period: Base Study (Cycle 1)
Arm/Group | Aprepitant Regimen | Control Regimen
Started | 155 | 152
Received Study Treatment | 152 | 150
Completed | 150 | 149
Not Completed | 5 | 3
Not completed — Adverse Event | 2 | 0
Not completed — Physician Decision | 0 | 1
Not completed — Protocol Violation | 2 | 0
Not completed — Withdrawal by Subject | 1 | 2
Period: Optional Extension (Cycles 2-6)
Arm/Group | Aprepitant Regimen | Control Regimen
Started | 171 | 0
Completed | 46 | 0
Not Completed | 125 | 0
Not completed — Adverse Event | 2 | 0
Not completed — Completed Chemotherapy Regimen | 51 | 0
Not completed — Did Not Meet Additional Criteria | 25 | 0
Not completed — Did Not Respond To Chemotherapy Regimen | 4 | 0
Not completed — Lack of Efficacy | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Physician Decision | 19 | 0
Not completed — Protocol Violation | 4 | 0
Not completed — Withdrawal by Subject | 18 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population: all randomized participants who received study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Aprepitant Regimen | Control Regimen | Total
Number analyzed (Participants) | 152 | 150 | 302
Age, Continuous [Mean (Standard Deviation); unit: Months] | 97.7 (63.2) | 99.4 (60.9) | 98.5 (62.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68 | 71 | 139
  Male | 84 | 79 | 163

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Complete Response in the Delayed Phase of Cycle 1
Description: Delayed Phase was defined as 25-120 hours after the start of chemotherapy. Complete response was defined as no vomiting or retching and no use of rescue medication in the delayed phase of Cycle 1.
Time Frame: 25 to 120 hours after the start of chemotherapy
Population: Intent-to-treat (ITT) population: all randomized participants who received study medication. Results for Cycles 2-6 were not included because this outcome measure is for Cycle 1 only.
Measure: Number; unit: Percentage of participants
Arm/Group | Aprepitant Regimen | Control Regimen
Number analyzed (Participants) | 152 | 150
Percentage of participants | 50.7 | 26.0
Statistical Analysis 1: Comparison: Aprepitant Regimen vs Control Regimen; Test type: Superiority or Other; p < 0.01, Cochran-Mantel-Haenszel; Stratified by age group, use of dexamethasone as an anti-emetic, and receipt of very high risk emetogenic chemotherapy

2. Secondary Outcome: Percentage of Participants With a Complete Response in the Acute Phase of Cycle 1
Description: Acute phase was defined as 0 to 24 hours after the start of chemotherapy. Complete response was defined as no vomiting or retching and no use of rescue medication in the acute phase of Cycle 1.
Time Frame: 0 to 24 hours after initiation of chemotherapy
Population: ITT population: all randomized participants who received study medication. Results for Cycles 2-6 were not included because this outcome measure is for Cycle 1 only.
Measure: Number; unit: Percentage of participants
Arm/Group | Aprepitant Regimen | Control Regimen
Number analyzed (Participants) | 152 | 150
Percentage of participants | 66.4 | 52.0
Statistical Analysis 1: Comparison: Aprepitant Regimen vs Control Regimen; Test type: Superiority or Other; p < 0.05, Cochran-Mantel-Haenszel; Stratified by age group, use of dexamethasone as an anti-emetic, and receipt of very high risk emetogenic chemotherapy

3. Secondary Outcome: Percentage of Participants With a Complete Response in the Overall Phase of Cycle 1
Description: Overall phase was defined as 0 to 120 hourse after the start of chemotherapy. Complete response was defined as no vomiting or retching and no use of rescue medication in the overall phase of Cycle 1.
Time Frame: 0 to 120 hours after initiation of chemotherapy
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Aprepitant Regimen | Control Regimen
Number analyzed (Participants) | 152 | 150
Percentage of participants | 40.1 | 20.0
Statistical Analysis 1: Comparison: Aprepitant Regimen vs Control Regimen; Test type: Superiority or Other; p < 0.01, Cochran-Mantel-Haenszel; Stratified by age group, use of dexamethasone as an anti-emetic, and receipt of very high risk emetogenic chemotherapy

4. Secondary Outcome: Percentage of Participants With No Vomiting in the Overall Phase of Cycle 1
Description: Overall phase was defined as 0 to 120 hourse after the start of chemotherapy. No vomiting was defined as no emesis or retching or dry heaves in the overall phase of Cycle 1.
Time Frame: 0 to 120 hours after initiation of chemotherapy
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Aprepitant Regimen | Control Regimen
Number analyzed (Participants) | 152 | 150
Percentage of participants | 46.7 | 21.3
Statistical Analysis 1: Comparison: Aprepitant Regimen vs Control Regimen; Test type: Superiority or Other; p < 0.01, Cochran-Mantel-Haenszel; Stratified by age group, use of dexamethasone as an anti-emetic, and receipt of very high risk emetogenic chemotherapy

ADVERSE EVENTS:
Description: Intent-to-treat (ITT) population: all randomized participants who received study medication.
Groups:
- Aprepitant Regimen Cycle 1: Participants 12 to 17 years of age, Day 1: aprepitant 125 mg capsule orally (PO) + ondansetron, Days 2 to 3: aprepitant 80 mg capsule PO. Participants 6 months to <12 years of age, Day 1: aprepitant powder for suspension (PFS), 3.0 mg/kg (up to 125 mg) + ondansetron, Days 2 to 3: aprepitant PFS, 2.0 mg/kg (up to 80 mg).
- Control Regimen Cycle 1: Participants 12 to 17 years of age, Day 1: matching placebo for aprepitant 125 mg capsule oral (PO) + ondansetron Days 2 to 3: matching placebo for aprepitant 80 mg capsule PO. Participants 6 months to <12 years of age, Day 1: matching placebo PFS: 3.0 mg/kg (up to 125 mg) + ondansetron, Days 2 to 3: matching placebo PFS: 2.0 mg/kg (up to 80 mg).
- Aprepitant Regimen Cycles 2-6: Participants completing Cycle 1 from either the aprepitant or the control regimen who meet eligibility criteria: Participants 12 to 17 years of age, Day 1: aprepitant 125 mg capsule orally (PO) + ondansetron, Days 2 to 3: aprepitant 80 mg capsule PO. Participants 6 months to <12 years of age, Day 1: aprepitant powder for suspension (PFS), 3.0 mg/kg (up to 125 mg) + ondansetron, Days 2 to 3: aprepitant PFS, 2.0 mg/kg (up to 80 mg).
Arm/Group | Aprepitant Regimen Cycle 1 | Control Regimen Cycle 1 | Aprepitant Regimen Cycles 2-6
Serious Adverse Events (participants affected / at risk) | 46/152 | 41/150 | 84/170
Other Adverse Events (participants affected / at risk) | 88/152 | 84/150 | 136/170
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aprepitant Regimen Cycle 1 (N=152) | Control Regimen Cycle 1 (N=150) | Aprepitant Regimen Cycles 2-6 (N=170)
Agranulocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 2 (2) | 3 (3) | 9 (11)
Bone marrow failure (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 23 (23) | 22 (22) | 53 (88)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 4 (4) | 0 (0) | 4 (6)
Pancytopenia (Blood and lymphatic system disorders) | 3 (3) | 6 (6) | 4 (7)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Caecitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Duodenitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastritis erosive (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2) | 3 (3) | 8 (9)
Catheter site pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (1)
Mucosal inflammation (General disorders) | 2 (2) | 2 (2) | 3 (3)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 2 (2) | 8 (8)
Thrombosis in device (General disorders) | 0 (0) | 0 (0) | 1 (1)
Hepatotoxicity (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Bacillus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Anaphylactic shock (Immune system disorders) | 1 (1) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Balanoposthitis infective (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Enterobiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Enterococcal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis clostridial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Otitis media acute (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Periorbital cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Postoperative wound infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Varicella (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Viral infetion (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2) | 3 (5)
Postoperative wound complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)
Drug clearance decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Electrocardiogram T wave inversion (Investigations) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 2 (2) | 4 (5)
Platelet count decreased (Investigations) | 2 (2) | 0 (0) | 1 (1)
White blood cell count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 4 (4)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Epithelioid sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Neuroblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Osteosarcoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Tumor haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Convulsion (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Renal tubular disorder (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Tracheal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aprepitant Regimen Cycle 1 (N=152) | Control Regimen Cycle 1 (N=150) | Aprepitant Regimen Cycles 2-6 (N=170)
Anaemia (Blood and lymphatic system disorders) | 24 (25) | 35 (38) | 62 (134)
Leukopenia (Blood and lymphatic system disorders) | 8 (9) | 10 (11) | 13 (22)
Neutropenia (Blood and lymphatic system disorders) | 17 (17) | 18 (20) | 39 (74)
Thrombocytopenia (Blood and lymphatic system disorders) | 15 (15) | 14 (16) | 38 (80)
Abdominal pain (Gastrointestinal disorders) | 11 (15) | 10 (15) | 17 (26)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 10 (12)
Constipation (Gastrointestinal disorders) | 3 (3) | 6 (6) | 12 (15)
Diarrhoea (Gastrointestinal disorders) | 8 (11) | 8 (8) | 16 (23)
Nausea (Gastrointestinal disorders) | 13 (20) | 17 (20) | 42 (78)
Stomatitis (Gastrointestinal disorders) | 5 (6) | 4 (4) | 12 (16)
Vomiiting (Gastrointestinal disorders) | 21 (31) | 20 (21) | 59 (152)
Mucosal inflammation (General disorders) | 1 (1) | 5 (5) | 11 (13)
Pyrexia (General disorders) | 8 (8) | 10 (10) | 22 (27)
Haemoglobin decreased (Investigations) | 8 (9) | 6 (7) | 14 (27)
Neutrophil count decreased (Investigations) | 12 (12) | 17 (19) | 32 (83)
Plastelet count decreased (Investigations) | 10 (10) | 15 (16) | 26 (58)
White blood cell count decreased (Investigations) | 5 (5) | 6 (6) | 12 (15)
Headache (Nervous system disorders) | 11 (11) | 7 (7) | 14 (15)
Cough (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 5 (6) | 18 (25)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3) | 10 (15)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 11 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission. Sponsor review can be expedited to meet publication timelines.